CLINICAL TRIAL: NCT07405463
Title: A Randomized, Double-Blind, Controlled Study of Transcranial Direct Current Stimulation Intervention on Fear Reversal in Patients With Anxiety Disorders
Brief Title: Effects of tDCS on Fear Reversal in Patients With Anxiety Disorders
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Jingchu Hu (Other)
Responsible Party: Sponsor-Investigator, Jingchu Hu, Dr. Jingchu Hu, Shenzhen Kangning Hospital
Organization: Shenzhen Kangning Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KN2025407
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Anxiety Disorders
Keywords: Transcranial Direct Current Stimulation; tDCS; Fear Reversal; Anxiety; Dorsolateral Prefrontal Cortex; Ventromedial Prefrontal Cortex; Cognitive Flexibility
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active Comparator: Cathodal rDLPFC (Experimental): Participants receive inhibitory stimulation over the right dorsolateral prefrontal cortex.
  Interventions: Device: Cathodal tDCS (rDLPFC)
- Active Comparator: Anodal vmPFC (Experimental): Participants receive excitatory stimulation over the ventromedial prefrontal cortex.
  Interventions: Device: Anodal tDCS (vmPFC)
- Sham Comparator: Sham tDCS (Sham Comparator): Participants receive a pseudo-stimulation that mimics the sensation of real tDCS but delivers no therapeutic current.
  Interventions: Device: Sham tDCS
- Active Comparator: Anodal lDLPFC (Active Comparator): Participants receive excitatory stimulation over the left dorsolateral prefrontal cortex (positive control).
  Interventions: Device: Anodal tDCS (lDLPFC)

INTERVENTIONS:
Device: Cathodal tDCS (rDLPFC) — Current intensity: 2.0 mA. Duration: 25 minutes. Cathode placed over F4 (10-20 system), Anode over contralateral deltoid.
  Arms: Active Comparator: Cathodal rDLPFC
Device: Anodal tDCS (vmPFC) — Current intensity: 2.0 mA. Duration: 25 minutes. Anode placed over Fpz (10-20 system), Cathode over Oz.
  Arms: Active Comparator: Anodal vmPFC
Device: Sham tDCS — Current ramps up for 30 seconds and then fades to zero to mimic skin sensation, with no sustained current for the rest of the 25 minutes.
  Arms: Sham Comparator: Sham tDCS
Device: Anodal tDCS (lDLPFC) — Current intensity: 2.0 mA. Duration: 25 minutes. Anode placed over F3 (10-20 system), Cathode over contralateral deltoid.
  Arms: Active Comparator: Anodal lDLPFC

SUMMARY:
This study evaluates the effects of single-session Transcranial Direct Current Stimulation (tDCS) on fear reversal learning in patients with anxiety disorders. Participants will be randomized into four groups to receive either active stimulation targeting specific brain regions (right DLPFC or vmPFC), an active control stimulation, or sham stimulation. The main goal is to determine if modulating these brain areas can improve the ability to update safety and threat associations.

DETAILED DESCRIPTION:
Anxiety disorders are characterized by deficits in fear regulation and cognitive flexibility, specifically the inability to inhibit fear responses when a threat becomes safe (fear reversal). Neurobiological models suggest this is linked to hyperactivity in the right dorsolateral prefrontal cortex (rDLPFC) and hypoactivity in the ventromedial prefrontal cortex (vmPFC).

This randomized, double-blind, sham-controlled study aims to verify if tDCS can improve fear reversal performance. The study involves 140 patients with anxiety disorders assigned to one of four arms:

Cathodal tDCS over the right DLPFC (inhibitory); Anodal tDCS over the vmPFC (excitatory); Sham tDCS (placebo); Anodal tDCS over the left DLPFC (active control). During the 25-minute stimulation session, participants will perform a computerized fear reversal task. Physiological data (Skin Conductance Response) and subjective anxiety ratings will be recorded simultaneously to assess the intervention's impact on cognitive and emotional regulation.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 60 years old. Right-handed. Meeting the DSM-5 diagnostic criteria for Gambling Disorder (GD). South Oaks Gambling Screen (SOGS) score ≥ 5. Normal or corrected-to-normal vision and hearing. Willingness to provide written informed consent and participate in the study.

Exclusion Criteria:

History of other severe psychiatric disorders (e.g., schizophrenia, bipolar disorder, severe depression) or neurological diseases (e.g., epilepsy, stroke, brain tumor).

History of substance abuse or dependence (excluding nicotine) in the past 6 months.

Current use of psychotropic medications that may affect cortical excitability (e.g., antidepressants, antipsychotics, anticonvulsants).

Presence of metallic implants in the head or neck area (e.g., cochlear implants, aneurysm clips) or cardiac pacemakers.

Skin lesions or sensitivity at the stimulation sites on the scalp. Pregnancy or lactation. Participation in other neuromodulation studies within the last 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 140 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Mean Accuracy Rate in the Reversal Phase of the Fear Reversal Task | During the intervention (Day 1, approximately 25 minutes)
  The percentage of correct responses during the reversal phase of the computerized task, where participants must inhibit previous fear associations and learn new safety signals. Higher scores indicate better cognitive flexibility.

SECONDARY OUTCOMES:
Reaction Time in the Reversal Phase | During the intervention (Day 1, approximately 25 minutes)
  The response time (in milliseconds) to the new CS+ (formerly CS-) and new CS- (formerly CS+) stimuli during the reversal phase.
Skin Conductance Response (SCR) Amplitude | During the intervention (Day 1, approximately 25 minutes)
  The amplitude of physiological skin conductance responses to Conditioned Stimuli (CS+ and CS-), serving as an objective measure of physiological arousal and fear response.
Subjective Anxiety Score (VAS) | During the intervention (Day 1, assessed intermittently during the 25-minute task)
  Self-reported anxiety levels measured using a Visual Analog Scale (VAS). Scores range from 0 (no anxiety) to 10 (extreme anxiety).

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Kangning Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No